CLINICAL TRIAL: NCT04073888
Title: Study of the Spermatic Characteristics of Patients With Fabry Disease
Acronym: FERTIFABRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2008/14
Record Dates: First submitted 2019-08-23; First posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): Men with Fabry Disease
  Interventions: Procedure: Semen collection

INTERVENTIONS:
Procedure: Semen collection — Semen collection for seminogram and spermocytogram

SUMMARY:
The objective of this project is to estimate the prevalence of spermatic abnormalities in patients with Fabry disease.The main objective of this project is to estimate the prevalence of spermatic abnormalities in patients with Fabry disease.

DETAILED DESCRIPTION:
Fabry disease is a lysosomal storage burden of X-linked genetic transmission due to alpha-galactosidase deficiency. This enzyme deficiency causes deposits of globotriaosylceramide in virtually all cell types of the body. The majority of hemizygous men develop a severe multisystemic disease dominated by renal failure, neurological and cardiac involvement. There is a specific treatment based on enzyme replacement therapy.

The incidence of Fabry disease is estimated between 1/60000 and 1/3500 in the general population.

Infertility in Fabry disease is poorly documented. Only a few cases have been reported, from alteration of spermogram to azoospermia. The identification of deposits suggestive of Gb3 in light microscopy and electron microscopy at the level of the genital tract argues in favor of the attack of this device. The low prevalence of Fabry disease requires a cross-sectional multicenter study to determine the frequency of alterations in sperm characteristics, their impact on fertility, and the possible effect of substitution therapy, in order to establish appropriate measures. adequate preventive measures.

The objective of this project is to estimate the prevalence of spermatic abnormalities in patients with Fabry disease.The main objective of this project is to estimate the prevalence of spermatic abnormalities in patients with Fabry disease.

ELIGIBILITY:
Inclusion Criteria:

* male patients with Fabry disease regardless of the clinical form of the disease; treated with enzyme replacement therapy or not (from the initial diagnosis). The definite diagnosis of Fabry disease will be established on the deficit of the activity of alpha galactosidase A (<12%). A molecular genetic study is desirable but not mandatory,
* patients aged 18 to 65,
* giving their free and informed consent to participate, after information on the research.

Exclusion Criteria:

* persons placed under the protection of justice,
* unaffiliated or non-beneficiary subject of a social security scheme.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Semen collection
Enrollment: 22 (Actual)
Dates: Start 2009-02-20 (Actual); Primary Completion 2013-10-18 (Actual); Study Completion 2013-10-18 (Actual)

PRIMARY OUTCOMES:
volume (ml) of sperm | At Day 1
  Spermogram characteristics
pH of sperm | At Day 1
  Spermogram characteristics
Count (million / ml) of spermatozoids | At Day 1
  Spermogram characteristics
Mobility (%) and mobility type of spermatozoa according to WHO classification of spermatozoids | At Day 1
  Spermogram characteristics
Total number of spermatozoa in one ejaculate | At Day 1
  Spermogram characteristics
Total number of progressive motile spermatozoa | At Day 1
  Spermogram characteristics
Existence of leukospermia yes/no | At Day 1
  Spermogram characteristics
% of typical forms of spermatozoids | At Day 1
  Characteristics of spermocytogram
Multiple Anomalies Index (MAI) of spermatozoids | At Day 1
  Characteristics of spermocytogram

CONTACTS AND LOCATIONS:
Overall Officials: Alice PAPAXANTHOS, Dr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No